CLINICAL TRIAL: NCT01609803
Title: Tissue Microarray Studies of the 12q13-q14 Amplicon in Alveolar Rhabdomyosarcoma
Brief Title: Studying Protein Expression in Tissue Samples From Younger Patients With Rhabdomyosarcoma
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: ARST12B7; NCI-2012-01972 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); COG-ARST12B7 (Other: Children's Oncology Group)
Record Dates: First submitted 2012-05-30; First posted 2012-06-01 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: Alveolar Childhood Rhabdomyosarcoma; Embryonal Childhood Rhabdomyosarcoma; Previously Treated Childhood Rhabdomyosarcoma; Previously Untreated Childhood Rhabdomyosarcoma; Recurrent Childhood Rhabdomyosarcoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — tissue samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Correlative studies: Formalin-fixed paraffin-embedded tissue samples are analyzed for 12q13-q14 frequency and protein overexpression by FISH and IHC.
  Interventions: Other: laboratory biomarker analysis

INTERVENTIONS:
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This research trial studies protein expression in tissue samples from younger patients with rhabdomyosarcoma. Studying samples of tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help doctors find better ways to treat cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To investigate (in two stages) which proteins are overexpressed in association with 12q13-q14 amplification by applying fluorescence in situ hybridization (FISH) and immunohistochemical (IHC) assays to a panel of alveolar rhabdomyosarcomas (ARMS) cases organized into tissue microarrays.

OUTLINE:

Formalin-fixed paraffin-embedded tissue samples are analyzed for 12q13-q14 frequency and protein overexpression by FISH and IHC.

ELIGIBILITY:
Inclusion Criteria:

* Slides of the 2006 alveolar rhabdomyosarcoma (ARMS) TMA and the 2009 ARMS/anaplastic embryonal rhabdomyosarcoma (ERMS) TMA

  * PAX3-FOXO1-positive tumors
  * PAX7-FOXO1-positive tumors
  * Fusion-negative tumors

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Tissue samples from younger patients with rhabdomyosarcoma from 2006
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2012-06; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Amplification and fusion status as a result of the 12q13-q14 amplification event | Baseline
  Fisher's exact test will be used. For a contingency table other than 2 x 2, the Freeman-Halton test (an extension of Fisher's exact test) will be applied instead.

CONTACTS AND LOCATIONS:
Overall Officials: Frederick Barr, MD, Principal Investigator — Children's Oncology Group
Locations (1):
- Children's Oncology Group, Monrovia, California, United States